CLINICAL TRIAL: NCT03751397
Title: Estimation of Kidney Function Through Combination of Renal Biomarkers in Blood and Urine of Healthy Infants and Children
Acronym: KidMaCare
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00884; ks18Pfister
Record Dates: First submitted 2018-11-13; First posted 2018-11-23 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Renal Biomarkers in Children
Keywords: Creatinine; Albumin; Cystatin C; Neutrophil gelatinase-associated lipocalin (NGAL); beta-trace Protein; beta-2 Microglobulin; Uromodulin
MeSH Terms: interventions — Hematologic Tests; Creatinine; Cystatin C; Lipocalin-2; prostaglandin R2 D-isomerase; beta 2-Microglobulin; Uromodulin; Urinalysis; Albumins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood test for renal biomarkers (creatinine, cystatin C, Neutrophil gelatinase-associated lipocalin, beta-trace protein, beta-2 microglobulin, uromodulin) — relationship between the different biomarkers by linear regression analysis is assessed; influence of demographic variables (age, body weight, body surface area) is investigated by multivariate regression.
Other: urine test for renal biomarkers (creatinine, cystatin C, Neutrophil gelatinase-associated lipocalin, beta-trace protein beta-2 microglobulin, uromodulin, albumin) — relationship between the different biomarkers by linear regression analysis is assessed; influence of demographic variables (age, body weight, body surface area) is investigated by multivariate regression.

SUMMARY:
To characterize the relationship of renal biomarkers (Creatinine, albumin, Cystatin C, NGAL, beta-trace protein, beta-2 microglobulin, and uromodulin) between each other and the variation over age, measured in serum and urine of healthy children. Unused residual blood and urine samples will be used for testing the renal Parameters.

DETAILED DESCRIPTION:
Despite relevant research in renal biomarkers, there is currently no optimal marker available that reliably quantifies kidney function and indicates kidney injury in its early stages. The combination of two or more biomarkers might be a more promising approach than investigating a single parameter. The relationship of renal biomarkers (creatinine, albumin, Cystatin C, NGAL, beta-trace protein, beta-2 microglobulin, and uromodulin) between each other and the variation over age in infants and children (without chronic kidney disease) is investigated.

The biomarkers in urine samples are explored to find less invasive means of quantifying renal health.

Patients between the age of 0 and 12 years undergoing blood with or without urine sampling as part of their diagnostic workup are eligible for the study. Unused residual blood and urine samples will be used for testing the renal parameters.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients for elective surgery, requiring venous access via peripheral venous canula

Exclusion Criteria:

* chronic kidney disease
* acute kidney failure (stage 2 or above as defined by Kidney Disease Improving Global Outcomes (KDIGO) consensus 2012))
* sepsis
* shock
* major haemorrhage
* second or third degree burns
* liver failure
* chronic diseases with effecting the kidney (systemic lupus erythematosus, amyloidosis)

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy patients between the age of 0 and 15 years visiting the Short Stay Unit of the University of Basel Children's Hospital for elective surgery and requiring venous access via peripheral venous canula are eligible for study participation
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Serum concentration of creatinine (ymol/l) | single point in time at subject enrollment
  blood test for renal biomarker
Serum concentration of cystatin C (mg/l) | single point in time at subject enrollment
  blood test for renal biomarker
Serum concentration of Neutrophil gelatinase-associated lipocalin (ng/ml) | single point in time at subject enrollment
  blood test for renal biomarker
Serum concentration of beta-trace Protein (mg/l) | single point in time at subject enrollment
  blood test for renal biomarker
Serum concentration of beta-2 Microglobulin (mg/l) | single point in time at subject enrollment
  blood test for renal biomarker
Serum concentration of Uromodulin (ng/ml) | single point in time at subject enrollment
  blood test for renal biomarker
Urine concentration of creatinine (mmols/kg/24h) | single point in time at subject enrollment
  Urine test for renal biomarker
Urine concentration of cystatin C (mg/l) | single point in time at subject enrollment
  Urine test for renal biomarker
Urine concentration of Neutrophil gelatinase-associated lipocalin (yg/l) | single point in time at subject enrollment
  Urine test for renal biomarker
Urine concentration of beta-trace Protein (mg/l) | single point in time at subject enrollment
  Urine test for renal biomarker
Urine concentration of beta-2 microglobulin (mg/l) | single point in time at subject enrollment
  Urine test for renal biomarker
Urine concentration of uromodulin (ng/ml) | at time of enrollment
  Urine test for renal biomarker
Urine concentration of Albumin (mg/l) | at time of enrollment
  Urine test for renal biomarker
Plasma protein binding of survival motor neuron (SMN) 2 splicing modifiers | single point in time at subject enrollment
  blood test for spinal muscular atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pfister, Prof. Dr. MD, Principal Investigator — University of Basel Children's Hospital
Locations (1):
- University of Basel Children's Hospital, Basel, Switzerland